CLINICAL TRIAL: NCT03374189
Title: Single Blind Randomized Control Trial Evaluating Efficacy and Safety of EZ-Close Port-site Closure Device Versus Carter-Thomason Device
Brief Title: Prospective Study on a Novel Port-site Closure Device (EZ Close): Effectiveness and Comparison With Carter-Thomason
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Principal Investigator, Hee Youn Kim, Assistant Professor, Saint Vincent's Hospital, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EZVSCT
Record Dates: First submitted 2017-12-11; First posted 2017-12-15 (Actual); Results first posted 2019-02-04 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Surgical Port Site Hernia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EZ Close arm (Experimental): EZ close used for port-site closure.
  Interventions: Device: EZ close
- Carter Thomason arm (Active Comparator): Carter Thomason used for port-site closure.
  Interventions: Device: Carter Thomason

INTERVENTIONS:
Device: EZ close — EZ close used.
  Arms: EZ Close arm
Device: Carter Thomason — Carter Thomason used.
  Arms: Carter Thomason arm

SUMMARY:
This study aims to evaluate the efficacy and safety of a novel port-site closure device (EZ Close) by comparing it with the Carter-Thomason device.

DETAILED DESCRIPTION:
Port-site closure is a critical procedure after every laparoscopic surgery. Complications such as visceral organ injury, port-site hernia, infection, ascitic fluid leakage may occur during and after the procedure. Many devices were developed and utilized for the procedure and Carter-Thomason is one of the most commonly used device and validated with several studies. This study aims to evaluate the efficacy and safety of a novel port-site closure device (EZ Close) by comparing it with the Carter-Thomason device.

ELIGIBILITY:
Inclusion Criteria:

* All patients with laparoscopic ports over 10mm

Exclusion Criteria:

* Patients with laparoscopic ports under 10mm
* Patients who refused the study
* Patients who received concurrent surgery for other reason

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hee Youn Kim, Principal Investigator — St Vincent's Hospital
Locations (1):
- St. Vincent's Hospital, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] del Junco M, Okhunov Z, Juncal S, Yoon R, Landman J. Evaluation of a novel trocar-site closure and comparison with a standard Carter-Thomason closure device. J Endourol. 2014 Jul;28(7):814-8. doi: 10.1089/end.2014.0069. Epub 2014 Apr 23. PMID 24588556
- [Background] Shetty A, Adiyat KT. Comparison between hand suture and Carter-Thomason needle closure of port sites in laparoscopy. Urol J. 2014 Sep 2;11(4):1768-71. PMID 25194073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients recruited between July 2017 and June 2018 at St. Vincent's Hospital.
Period: Overall Study
Arm/Group | EZ Close Arm | Carter Thomason Arm
Started | 40 | 39
Completed | 39 | 39
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EZ Close Arm | Carter Thomason Arm | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (10.0) | 58.8 (16.2) | 62.1 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 31 | 28 | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 23.2 (2.8) | 23.6 (3.1) | 23.4 (2.9)
Operation time [Mean (Standard Deviation); unit: minutes] | 211.7 (90.0) | 217.3 (77.6) | 214.5 (83.6)
Operation type [Count of Participants; unit: Participants]
  Laparoscopic radical nephrectomy | 4 | 6 | 10
  Laparoscopic partial nephrectomy | 1 | 1 | 2
  Laparoscopic radical prostatectomy | 4 | 5 | 9
  Laparoscopic radical cystectomy | 2 | 3 | 5
  Robot-assisted radical nephrectomy | 0 | 1 | 1
  Robot-assisted partial nephrectomy | 8 | 8 | 16
  Robot-assisted radical prostatectomy | 16 | 10 | 26
  Robot-assisted radical cystectomy | 2 | 1 | 3
  Others | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Time Taken to Complete Closure
Description: The start of the procedure was defined as the point when the device was first inserted through the port-site and the end of the procedure was defined as the point when the port-site was removed from the port-site. A stopwatch was used to measure the time.
Time Frame: At the time of surgery
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | EZ Close Arm | Carter Thomason Arm
Number analyzed (Participants) | 39 | 39
seconds | 36.8 (10.1) | 48.9 (21.5)

2. Secondary Outcome: Number of Participants With Visceral Organ Injury
Description: Any inadvertent injury to organs or bleeding during procedure.
Time Frame: At the time of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | EZ Close Arm | Carter Thomason Arm
Number analyzed (Participants) | 39 | 39
Participants | 0 | 0

3. Secondary Outcome: Number of Participants With Need for Additional Instrument
Description: Need for additional instrument during procedure
Time Frame: At the time of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | EZ Close Arm | Carter Thomason Arm
Number analyzed (Participants) | 39 | 39
Participants | 0 | 33

4. Secondary Outcome: Number of Participants With Port-site Hernia
Description: Herniation of bowel segments through port-site
Time Frame: 3 days post-op and within one months of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | EZ Close Arm | Carter Thomason Arm
Number analyzed (Participants) | 39 | 39
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Port-site Infection
Description: Redness, purulent discharge, tenderness at port-site
Time Frame: 3 days post-op and within one months of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | EZ Close Arm | Carter Thomason Arm
Number analyzed (Participants) | 39 | 39
Participants | 1 | 2

6. Secondary Outcome: Number of Participants With Ascitic Fluid Leakage
Description: Non-infective fluid leakage
Time Frame: 3 days post-op and within one months of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | EZ Close Arm | Carter Thomason Arm
Number analyzed (Participants) | 39 | 39
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Wound Dehiscence
Description: Wound dehiscence that required further treatment
Time Frame: 3 days post-op and within one months of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | EZ Close Arm | Carter Thomason Arm
Number analyzed (Participants) | 39 | 39
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Any adverse events other than the primary and secondary outcome measures were recorded during the study period. (At the time of the surgery, 3-days post-op and within 1 months of operation)
Arm/Group | EZ Close Arm | Carter Thomason Arm
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT03374189/Prot_SAP_000.pdf